CLINICAL TRIAL: NCT05904327
Title: The Use of Circulating Biomarkers in Oropharyngeal Cancer and Unknown Primary of Head and Neck - a Prospective Multicenter Study for Treatment Evaluation and Surveillance
Brief Title: Circulating Biomarkers in Oropharyngeal Cancers
Acronym: CIRCOS
Status: Active, not recruiting | Type: Observational
Sponsor: Region Örebro County (Other)
Collaborators: Region Stockholm (Other Government); Region Västmanland (Other); Dalarna County Council, Sweden (Other); Sormland County Council, Sweden (Other); Värmland County Council, Sweden (Other Government)
Responsible Party: Sponsor
Other Study IDs: 278627
Record Dates: First submitted 2023-04-17; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-04

CONDITIONS: Oropharynx Squamous Cell Carcinoma; Oropharynx Cancer; Tonsillar Cancer; Base of the Tongue Carcinoma
Keywords: circulating tumor DNA; HPV; human papilloma virus
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms; Tonsillar Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational longitudinal study is to learn about circulating tumor Human Papilloma Virus-DNA (ctHPV-DNA) as a biomarker for HPV positive oropharyngeal cancer and cancer of unknown primary of the head and neck. The main questions it aims to answer are:

* Can ctHPV-DNA be used for treatment evaluation in HPV positive oropharyngeal cancer and cancer of unknown primary of the head and neck?
* Can circulating HPV-DNA be used as a biomarker for recurrent disease during surveillance?

Participants will be asked to leave plasma samples at diagnose, at the end of treatment and at every clinical follow-up.

The patients are there own controls.

DETAILED DESCRIPTION:
In the multicenter study of CIRCOS, Circulating biomarkers in oropharyngeal cancer, patients with oropharyngeal cancer or cancer of unknown primary of the head and neck are consecutively included. Plasma samples are collected at diagnosis, at the end of treatment and during surveillance after treatment.

At diagnose participants will fill in informed consent and a form regarding known risk factors for cancer. Tissue from the tumor will be analyzed for HPV genotype with a multiplex q-PCR. Information about p16 will be collected from medical records.

ctHPV-DNA are short DNA fragments that leaks into the blood stream from tumor cells during apoptosis and necrosis. In the study, ctHPV-DNA will be extracted from blood plasma. Levels of ctHPV-DNA (copies/mL) will be measured using digital droplet PCR (ddPCR) with genotype specific assays (based on the result of q-PCR at diagnose) used in singleplex (SAGA diagnostics). A negative sample after treatment will be defined as a good molecular response for evaluation after treatment. Two consecutive, positive samples during surveillance will be defined as molecular recurrence. If a molecular recurrence is seen patients will be contacted and offered an extra clinical control at an Ear nose and throat department.

If a patient is HPV negative in tissue, the tissue will be analyzed with whole genome sequencing. If a mutation is found, a personalized ddPCR-kit will be used for plasma.

All patients will be followed for five years.

ELIGIBILITY:
Inclusion Criteria:

* Oropharyngeal cancer
* Cancer of unknown primary in the head and neck

Exclusion Criteria:

* Previous treatment of cancer in the oropharynx.
* Previous treatment of unknown primary tumor.
* Remote metastases
* Patients unwilling or unable to comply with the study protocol and follow-up schedule

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants are recruited from multidisciplinary conferences of head and neck cancer at Örebro University hospital - Region Örebro County, Västmanland's hospital - Region Västmanland and Karolinska University hospital - Region Stockholm. Örebro University hospital is a tertiary referral hospital of three regions in central Sweden (Region Värmland, Region Sörmland and Region Dalarna) and therefore patients from these regions will also be included in this study. All patients with OPSCC at any of the study centers will be asked to participate in CIRCOS. All study participants will sign an informed written consent upon inclusion
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
The accuracy of ctHPV-DNA as a biomarker for recurrent disease, measured in PPV and NPV | 5 year follow-up
  ctHPV-DNA will be evaluated by ddPCR. Two consecutive positive values will be defined as a molecular recurrance. The accuracy of the test will be presented with negative predictive value (NPV) and positive predictive value (PPV) at one, two (interim analysis) and at five year follow-up

SECONDARY OUTCOMES:
The correlation between molecular tumor burden (copies/mL) and radiological tumor burden (diameter and volume) using Kendall rank correlation coefficient. | 3 months follow-up
  Correlation of ctHPV-DNA and radiologic tumor burden at diagnosis and post treatment. ctHPV-DNA will be evaluated by ddPCR (copies/mL) at diagnose and at the end of treatment. The levels of ctHPV-DNA will be used as a measure of molecular tumor burden. The molecular tumor burden will be compared with the radiologic tumor burden, measured in diameter and volume in the diagnostic and evaluation computed tomography. The correlation will be calculated using Kendall rank correlation coefficient
A comparison between molecular (copies/mL) and radiological response to treatment according to RECIST (Response Evaluation Criteria in Solid Tumors) using Kruskal wallis test. | 3 months follow-up
  The kinetics in ctHPV-DNA and will be compared to radiological confirmed treatment response in order to test ctHPV-DNA as a biomarker for treatment response. Radiological response will be evaluated according to the RECIST-criteria. Kinetics of ctHPV-DNA will be described as percentage change between pre- and post-treatment levels of ctHPV-DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Helenius, Study Director — Örebro University, Sweden
Locations (1):
- Anna Oldaeus Almerén, Örebro, Sweden

REFERENCES:
- [Derived] Almeren AO, Waenerlund M, Landstrom F, von Beckerath M, Qvick A, Carlsson J, Helenius G. Circulating Tumour DNA as a Complementary Tool for Treatment Evaluation in HPV-Associated Head and Neck Squamous Cell Carcinoma: An Observational Cohort Study. Clin Otolaryngol. 2025 Sep;50(5):831-839. doi: 10.1111/coa.14317. Epub 2025 Apr 22. PMID 40260766
- [Derived] Qvick A, Andersson E, Oldaeus Almeren A, Waenerlund M, Stenmark B, Karlsson C, Karlsson MG, Helenius G. Sensitive and Specific Droplet Digital PCR Assays for Circulating Tumor HPV DNA: Development, Validation, and Clinical Application in HPV-Associated Cancers. Mol Diagn Ther. 2024 Nov;28(6):835-845. doi: 10.1007/s40291-024-00743-9. Epub 2024 Sep 26. PMID 39325260